CLINICAL TRIAL: NCT04787458
Title: Effect of Abdominal Binder After Laparoscopic Cholecystectomy on Enhanced Recovery(ABC) : a Randomized Controlled Trial
Brief Title: Effect of Abdominal Binder After Laparoscopic Cholecystectomy on Enhanced Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Sung Ryol Lee, Hepato-biliary and pancreatic department of General Surgery, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002041
Record Dates: First submitted 2021-02-09; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In subjects allocated to the abdominal binder group, the abdomen binder with a standard height of 22 cm (Sejung Korea, Seoul, Republic of Korea) was applied before leaving the operating room. Subjects were carefully instructed to use the abdominal binder during at least the first 2 consecutive days and night, and to reposition the abdominal binder correctly when needed.
  Interventions: Device: abdomen binder (Sejung Korea, Seoul, Republic of Korea)
- Control group (No Intervention): subjects allocated in the control group, subjects were not given any opportunity to ware an abdominal binder.

INTERVENTIONS:
Device: abdomen binder (Sejung Korea, Seoul, Republic of Korea) — abdomen binder with a standard height of 22 cm (Sejung Korea, Seoul, Republic of Korea)
  Arms: Experimental group

SUMMARY:
There have been reports that abdominal binder use after laparoscopic or open surgery affects postoperative respiratory function, walking performance, and pain but no study has evaluated binder use solely for laparoscopic cholecystectomy surgery. Therefore, the investigators performed a randomized controlled trial to evaluate the effect of abdominal binders after laparoscopic cholecystectomy by comparing postoperative outcomes in two patient groups.

DETAILED DESCRIPTION:
Abdominal binders help to prevent postoperative complications, however, their use is controversial because of a lack of evidence for their effectiveness and because they also confer disadvantages. The purpose of this randomized controlled trial was to compare the effects of abdominal binder after laparoscopic cholecystectomy on pain, degree of comfort, time until ambulation, walking ability, return of bowel function, and diet resumption.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* American Society of Anesthesiologists Physical Status classification I and II

Exclusion Criteria:

* history of ventral hernia
* walking disability
* chronic obstructive respiratory disease
* malignancy
* chronic pain syndrome
* open conversion
* inability to complete the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-08-09 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
degree of comfort | Until dischage, an average of 2.5 days
  Questionnaire response options ranged from very comfortable (5) to very Questionnaire response options ranged from very comfortable (5) to very uncomfortable (0).
postoperative pain | 12 hours after surgery
  Subjects rated postoperative pain intensity using a visual analog scale (0-10, VAS) at 12 hours after surgery
postoperative pain | 24 hours after surgery
  Subjects rated postoperative pain intensity using a visual analog scale (0-10, VAS) at 24 hours after surgery
postoperative pain | 48 hours after surgery
  Subjects rated postoperative pain intensity using a visual analog scale (0-10, VAS) at 48 hours after surgery

SECONDARY OUTCOMES:
Postoperative hospital stay | Until dischage, an average of 2.3 days
  Postoperative hospital stay days to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No